CLINICAL TRIAL: NCT02024529
Title: A Phase 3 Randomized, Placebo-controlled, Double-blind Study to Evaluate the Safety and Efficacy of a Single Intra-articular Injection of Ampion in Adults With Pain Due to Osteoarthritis (OA) of the Knee
Brief Title: A Randomized, Controlled Study to Evaluate Efficacy and Safety of Intra-articular Ampion for Osteoarthritis Pain in Knee
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ampio Pharmaceuticals. Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AP-004-A
Record Dates: First submitted 2013-12-26; First posted 2013-12-31 (Estimated); Results first posted 2022-08-09 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2022-07

CONDITIONS: Osteoarthritis of the Knee
Keywords: Osteoarthritis; osteoarthritis of the knee
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AMPION™ 4 mL dose (Experimental): 4 mL injection of Ampion
  Interventions: Biological: 4 mL injection of Ampion
- Placebo 4 mL dose (Placebo Comparator): 4 mL injection of placebo
  Interventions: Drug: 4 mL Injection of Placebo

INTERVENTIONS:
Biological: 4 mL injection of Ampion — 4 mL injection of Ampion
  Arms: AMPION™ 4 mL dose
Drug: 4 mL Injection of Placebo — 4 mL Injection of Placebo
  Other Names: Saline
  Arms: Placebo 4 mL dose

SUMMARY:
This study will evaluate the efficacy of an Intra-Articular Injection of Ampion™ in Adults with pain due to osteoarthritis of the knee.

DETAILED DESCRIPTION:
A Randomized, Placebo-controlled, Double-Blind Study to Evaluate the Efficacy and Safety of an Intra-Articular Injection of Ampion™ in Adults with pain due to osteoarthritis of the knee.

The primary study objective was to evaluate the efficacy of 4 mL Ampion versus 4 mL saline intra-articular (IA) injection in treating knee pain when administered to subjects suffering from osteoarthritis (OA) of the knee (OAK).

The secondary study objectives included evaluation of the safety of an IA injection of Ampion vs saline, efficacy of IA injection of Ampion vs saline in improving knee function.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 35 years to 85 years old (inclusive) who are ambulatory but suffering from moderate to moderately severe pain from osteoarthritis in the index knee as evidenced by a rating of at least 1.5 on the WOMAC Index 3.1 5-point Likert Pain Subscale at screening.
2. Index knee must be symptomatic for greater than 6 months with a clinical diagnosis of OA and supported by radiological evidence (Kellgren Lawrence Grade II, III, IV). Confirmatory x-ray must be taken at Screening and assessed using Kellgren Lawrence grading system.
3. Moderate to moderately-severe OA pain in the index knee even with dosing of nonsteroidal anti-inflammatory drug (NSAID) in the 4 weeks prior to screening.
4. No analgesia (including acetaminophen [paracetamol]) taken 12 hours prior to an efficacy measure; and,
5. Able to provide written informed consent to participate in the study.
6. Willing and able to comply with all study requirements and instructions of the site study staff.

Exclusion Criteria:

1. Previous participation in an Ampion™ study.
2. Inflammatory or crystal arthropathies, acute fractures, history of aseptic necrosis or joint replacement in the affected knee, as assessed locally by the principal investigator.
3. Isolated patella femoral syndrome, also known as chondromalacia.
4. Any other disease or condition interfering with the free use and evaluation of the index knee for the duration of the trial (e.g., cancer, congenital defects, spine OA).
5. Major injury to the index knee within the 12 months prior to screening.
6. Severe hip OA ipsilateral to the index knee.
7. Presence of tense effusions.
8. Any pain that could interfere with the assessment of index knee pain (e.g., pain in any other part of the lower extremities, pain radiating to the knee).
9. Initiation or change in any pharmacological or non-pharmacological treatment for OA during the 4 weeks prior to randomization or likely to be changed during the duration of the study.
10. Use of the following medications anticipated to be required during the study:

    * Intra-articular pain medications in the study knee
    * Analgesics containing opioids. (NSAIDs may be continued at levels preceding the study and acetaminophen is available as a rescue medication during the study from the provided supply.)
    * Topical treatment on osteoarthritis index knee needed during the study
    * Use of significant anticoagulant therapy, oral or injectable, during the study (aspirin and clopidogrel are allowed)
    * Systemic treatments that may interfere with safety or efficacy assessments during the study such as immunosuppressants
11. Use of corticosteroids >10 mg prednisolone equivalent per day (if ≤10 mg prednisolone, the dose must be stable).
12. Use of human albumin treatment in the 3 months before randomization.
13. A history of allergic reactions to human albumin (reaction to non-human albumin such as egg albumin is not an exclusion criterion).
14. A history of allergic reactions to excipients in 5% human albumin (N-acetyltryptophan, sodium caprylate).
15. Principal Investigator considers the patient unfit for the study based on medical review and screening.

Ages: 35 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 538 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2014-05 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Howard Levy, MD, Study Director — Ampio Pharmaceuticals. Inc.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Cole B, McGrath B, Salottolo K, Bar-Or D. LMWF-5A for the Treatment of Severe Osteoarthritis of the Knee: Integrated Analysis of Safety and Efficacy. Orthopedics. 2018 Jan 1;41(1):e77-e83. doi: 10.3928/01477447-20171114-05. Epub 2017 Nov 21. PMID 29156068

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment of subjects occurred in medical clinics during the months of January and February 2014.
Pre-assignment Details: No pharmacological or non-pharmacological treatment targeting osteoarthritis (OA) started or changed during the 4 weeks prior to randomization or likely to be changed during the duration of the study.
Groups:
- Ampion 4 mL Injection: 4 mL Intra-articular injection of Ampion
- Placebo 4 mL Injection: 4 mL placebo intra-articular injection
  Placebo: Saline
Period: Overall Study
Arm/Group | Ampion 4 mL Injection | Placebo 4 mL Injection
Started | 269 | 269
Completed | 256 | 244
Not Completed | 13 | 25
Not completed — Withdrawal by Subject | 11 | 21
Not completed — Lost to Follow-up | 2 | 4

BASELINE CHARACTERISTICS:
Groups:
- Placebo 4 mL Injection: 4 mL placebo intra-articular injection
- Total: Total of all reporting groups
Arm/Group | Ampion 4 mL Injection | Placebo 4 mL Injection | Total
Number analyzed (Participants) | 269 | 269 | 538
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.1 (9.5) | 61.2 (9.6) | 60.6 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 151 | 159 | 310
  Male | 118 | 110 | 228
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 16 | 18 | 34
  Not Hispanic or Latino | 253 | 251 | 504
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 0 | 3
  Asian | 4 | 7 | 11
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 48 | 35 | 83
  White | 214 | 219 | 433
  More than one race | 0 | 5 | 5
  Unknown or Not Reported | 0 | 3 | 3
Region of Enrollment [Number; unit: participants]
  United States | 269 | 269 | 538
Weight (kg) [Mean (Standard Deviation); unit: kg] | 96.1 (24.0) | 95.1 (21.9) | 95.6 (23.0)
BMI (kg/m^2) [Mean (Standard Deviation); unit: kg/m^2] | 34.2 (8.1) | 34.2 (7.6) | 34.2 (7.9)
Kellgren-Lawrence (KL) Grade [Count of Participants; unit: Participants] — Kellgren-Lawrence grading is based on the radiologic features of osteoarthritis.
  Ann Rheum Dis. 1957;16:494-502.
  Grade II (Mild): Definite osteophytes, possible joint space narrowing.
  Grade III (Moderate): Moderate osteophytes, definite joint space narrowing, some sclerosis, possible bone-end deformity.
  Grade IV (Severe): Large osteophytes, marked joint space narrowing, severe sclerosis, definite bone-end deformity.
  Participants
    Kellgren-Lawrence Grade II | 67 | 66 | 133
    Kellgren-Lawrence Grade III | 105 | 90 | 195
    Kellgren-Lawrence Grade IV | 97 | 113 | 210
WOMAC Pain [Mean (Standard Deviation); unit: score on a scale] — The Western Ontario and McMaster Universities Arthritis Index (WOMAC) 3.1 evaluates Pain (5 items): during walking, using stairs, in bed, sitting or lying, and standing upright.
  Subjects respond to each subscale by using a 5-point Likert score. (0=none; 1=mild; 2=moderate; 3=severe; 4=extreme). Mean of the 5 scores constitutes the Baseline Pain Score.
  Higher scores are indicative of higher levels of self-reported pain.
  score on a scale | 2.38 (0.56) | 2.38 (0.58) | 2.38 (0.57)
WOMAC Function [Mean (Standard Deviation); unit: score on a scale] — WOMAC 3.1 evaluates Physical Function (17 items): using stairs, rising from sitting, standing, bending, walking, getting in/out of a car, shopping, putting on / taking off socks, rising from bed, lying in bed, getting in/out of bath, sitting, getting on/off toilet, heavy/light domestic duties.
  Subjects respond to each subscale by using a 5-point Likert score. (0=none; 1=mild; 2=moderate; 3=severe; 4=extreme). Mean of the 17 scores constitutes the Baseline Function Score.
  Higher scores are indicative of higher levels of limitations of self-reported physical function
  score on a scale | 2.45 (0.60) | 2.41 (0.63) | 2.43 (0.61)

OUTCOME MEASURES:

1. Primary Outcome: Change in WOMAC A Pain
Description: Mean Change in WOMAC A Pain (Western Ontario and McMaster Universities Arthritis Index) score from Baseline to 12 weeks. 5-point Likert scale (0=none to 4=extreme). A negative difference constitutes a decrease in pain with a greater negative value indicating a greater reduction in pain.
Time Frame: Scored at Baseline and 12 weeks
Population: Intent to Treat (ITT)
Measure: Mean (95% Confidence Interval); unit: score on a scale
Groups:
- Ampion 4 mL Injection: 4 mL Intra-articular injection of Ampion
  Ampion: <5 kiloDalton (kDa) ultrafiltrate of 5% human serum albumin
Arm/Group | Ampion 4 mL Injection | Placebo 4 mL Injection
Number analyzed (Participants) | 269 | 269
score on a scale | -0.81 [-0.91 to -0.71] | -0.81 [-0.91 to -0.70]
Statistical Analysis 1: Comparison: Ampion 4 mL Injection vs Placebo 4 mL Injection; Test type: Superiority; p = 0.97, ANCOVA — Adjusted for baseline WOMAC score

2. Secondary Outcome: Change in WOMAC C Function
Description: Mean change in WOMAC C function score (Western Ontario and McMaster Universities Arthritis Index) from Baseline to 12 weeks. 5-point Likert scale indicating limitation of function (0=none to 4=extreme). A greater negative value indicates a improvement in function.
Time Frame: Scored at Baseline and 12 weeks.
Population: Intent to Treat (ITT)
Measure: Mean (95% Confidence Interval); unit: score on a scale
Groups:
- Ampion 4 mL Injection: 4 mL Intra-articular injection of Ampion
  Ampion: <5 kDa ultrafiltrate of 5% human serum albumin
Arm/Group | Ampion 4 mL Injection | Placebo 4 mL Injection
Number analyzed (Participants) | 269 | 269
score on a scale | -0.76 [-0.87 to -0.66] | -0.77 [-0.88 to -0.67]
Statistical Analysis 1: Comparison: Ampion 4 mL Injection vs Placebo 4 mL Injection; Test type: Superiority; p = 0.75, ANCOVA — Adjusted for baseline WOMAC score

3. Post Hoc Outcome: Change in WOMAC A Pain of KL Grade IV Subset
Description: as for outcome 1
Time Frame: Scored at Baseline and 12 weeks
Population: Intent to Treat (ITT)
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Ampion 4 mL Injection | Placebo 4 mL Injection
Number analyzed (Participants) | 97 | 113
score on a scale | -0.82 [-0.99 to -0.66] | -0.65 [-0.81 to -0.49]
Statistical Analysis 1: Comparison: Ampion 4 mL Injection vs Placebo 4 mL Injection; Test type: Superiority; p = 0.18, ANCOVA; Adjusted for baseline WOMAC Score

4. Post Hoc Outcome: Change in WOMAC C Function of KL Grade IV Subset
Description: as for outcome 2
Time Frame: Scored at Baseline and 12 Weeks
Population: Intent to Treat (ITT)
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Ampion 4 mL Injection | Placebo 4 mL Injection
Number analyzed (Participants) | 97 | 113
score on a scale | -0.73 [-0.91 to -0.56] | -0.69 [-0.85 to -0.52]
Statistical Analysis 1: Comparison: Ampion 4 mL Injection vs Placebo 4 mL Injection; Test type: Superiority; p = 0.81, ANCOVA; Adjusted for baseline WOMAC Score

ADVERSE EVENTS:
Time Frame: 12 Weeks
Description: Patients will be followed for the occurrence of Adverse Events until 12 weeks after the first dose of study medication.
Groups:
- Ampion 4 mL Injection: 4 mL Intra-articular injection of Ampion
  Ampion: kDa ultrafiltrate of 5% human serum albumin
Arm/Group | Ampion 4 mL Injection | Placebo 4 mL Injection
All-Cause Mortality (participants affected / at risk) | 0/269 | 0/269
Serious Adverse Events (participants affected / at risk) | 6/269 | 4/269
Other Adverse Events (participants affected / at risk) | 65/269 | 71/269
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ampion 4 mL Injection (N=269) | Placebo 4 mL Injection (N=269)
Atrial Fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 3 (3) | 0 (0)
Hip Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Adenocarcinoma of Colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Non-Hodgkin's Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Ovarian Cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ampion 4 mL Injection (N=269) | Placebo 4 mL Injection (N=269)
Arthralgia (Musculoskeletal and connective tissue disorders) | 35 | 30
Upper Respiratory Tract Infection (Infections and infestations) | 7 | 11
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 6 | 4
Sinusitis (Infections and infestations) | 4 | 6
Fall (Injury, poisoning and procedural complications) | 5 | 4
Injection Site Pain (General disorders) | 4 | 5
Bronchitis (Infections and infestations) | 3 | 5
Contusion (Injury, poisoning and procedural complications) | 1 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes